CLINICAL TRIAL: NCT05149794
Title: Effects Of Calisthenic Exercises On Physical Fitness Among School Going Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/0766 Faseeh Zulqernain
Record Dates: First submitted 2021-09-23; First posted 2021-12-08 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Healthy Life Style; Physical Fitness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calisthenic Exercises (Experimental): The participants of this group perform calisthenic exercises.
  Interventions: Other: Calisthenic Exercises
- Conventional Training (No Intervention): The participants of this group perform activities of daily routines like playing cricket, taking swings etc

INTERVENTIONS:
Other: Calisthenic Exercises — Bunny Jumps, Bear Crawls, Bear Crawls, Bird Dog . these intervention were used
  Other Names: Calisthenic Exercises (Animal Style)
  Arms: Calisthenic Exercises

SUMMARY:
The study will be conducted to determine the effects of Calisthenic Exercise on Physical fitness among school going children .

DETAILED DESCRIPTION:
Callisthenic Exercises has proven effective in gaining strength, endurance and balance in adults and children age (11 to 17 years) but still evidence is less as compared to children age (8 to 13 years). calesthenics can be perform in door so for children who mostly stay t home or on gadget if perform these activities may improve their physical fitness

ELIGIBILITY:
Inclusion Criteria:

* Male school going children (8-13 year of age)
* Participants who are able to perform 11-12 repetitions of Calisthenic Exercises mentioned in my Study.
* BMI of school going children (8-13 year of age)

Exclusion Criteria:

* • Children with any disability.

  * Children with any acute illness.
  * History of any fracture.

Ages: 8 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Euro fit Fitness Testing Battery | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No